CLINICAL TRIAL: NCT02928575
Title: A Phase II Trial of Concurrent Sunitinib, Temozolomide and Radiation Therapy Followed by Adjuvant Temozolomide for Newly Diagnosed Glioblastoma Patients With an Unmethylated MGMT Gene Promoter
Brief Title: Combining Sunitinib, Temozolomide and Radiation to Treat Patients Diagnosed With Glioblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bassam Abdulkarim (Other)
Collaborators: Pfizer (Industry); Canadian Cancer Society (CCS) (Other)
Responsible Party: Sponsor-Investigator, Bassam Abdulkarim, PhD, MD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: McG 1132
Record Dates: First submitted 2016-01-14; First posted 2016-10-10 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma; Sunitinib; Temozolomide; Radiation Therapy,; MGMT; Biomarkers
MeSH Terms: conditions — Glioblastoma | interventions — Sunitinib; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunitinib, Temozolomide and Radiation Therapy (Experimental): Before concurrent treatment, patients will receive sunitinib orally at a dose of 12.5 mg once daily for one week prior to radiation. Patients will then receive a concomitant treatment of sunitinib at a dose of 12.5 mg once daily along with temozolomide (75 mg/m2 daily) along with radiotherapy (60 Gy in 30 fractions) over a period of 6 weeks. This concurrent treatment of sunitinib, temozolomide and radiotherapy is followed by a 1 month break after which the adjuvant temozolomide treatment is administered at a dose of 150/200mg/m2 daily, for 5 of 28 days over a period of 6 months.
  Interventions: Drug: Sunitinib; Drug: Temozolomide; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Sunitinib — Before concurrent treatment, patients will receive sunitinib orally at a dose of 12.5 mg once daily for one week prior to radiation. Patients will then receive a concomitant treatment of sunitinib at a dose of 12.5 mg once daily along with temozolomide (75 mg/m2 daily) along with radiotherapy (60 Gy in 30 fractions) over a period of 6 weeks.
  Other Names: Sutent (SU11248)
Drug: Temozolomide — Temozolomide (75 mg/m2 daily) will be administered along with sunitinib (12.5 mg once daily) and radiotherapy (60 Gy in 30 fractions) over a period of 6 weeks. This concurrent treatment of sunitinib, temozolomide and radiotherapy is followed by a 1 month break after which the adjuvant temozolomide treatment is administered at a dose of 150/200mg/m2 daily, for 5 of 28 days over a period of 6 months.
Radiation: Radiation Therapy — Patients will receive a concomitant treatment of radiotherapy (60 Gy in 30 fractions), sunitinib (12.5 mg once daily) and temozolomide (75 mg/m2 daily) over a period of 6 weeks.

SUMMARY:
The purpose of this study is to determine whether a combination of Sunitinib, Temozolomide and Radiation Therapy would be effective in the treatment of newly diagnosed Glioblastoma patients harboring tumors with unmethylated MGMT promoter.

DETAILED DESCRIPTION:
Glioblastoma multiforme (GBM), the most common primary brain tumor in adults is known for its highly invasive and angiogenic profile. Despite advances in different modalities of GBM treatment, the overall prognosis of GBM remains dismal. The current standard of care is Radiation Therapy (RT) at a dose of 60 Gy (30 fractions) for 6 weeks with concurrent Temozolomide (TMZ; 75 mg/m2 daily for 6 weeks) followed by adjuvant TMZ (150/200mg/m2 daily, for 5 of 28 days x 6 months). The DNA repair protein O6-methylguanine methyltransferase (MGMT) removes alkyl adducts at the O6 position of guanine and therefore counteracts the cytotoxic effects of alkylating agents such as TMZ. Thus, GBM patients harboring tumors with unmethylated MGMT promoter and increased MGMT protein expression do not derive benefit from TMZ treatment.

Sunitinib (Sutent, SU11248) is an oral multitargeted receptor tyrosine kinase (RTK) inhibitor with anti-angiogenic activities. Sunitinib has been approved by the FDA for the treatment of patients with gastrointestinal stromal tumors after disease progression on or intolerance to imatinib, for the treatment of patients with advanced renal cell carcinoma and for the treatment of patients with unresectable, locally advanced, or metastatic well-differentiated pancreatic neuroendocrine tumors (pNET). Previous pre-clinical data showed the efficacy of sunitinib in GBM. The investigators preclinical data highlighted the differential effect of sunitinib in GBM MGMT-positive tumors with a greater response to sunitinib in combination with RT and TMZ compared to MGMT-negative tumors.

In this phase II trial, Investigator will test the efficacy and the safety of combining Sunitinib with RT and TMZ in newly diagnosed GBM patients displaying tumors with unmethylated MGMT promoter. Based on the investigators preclinical findings, patients with MGMT (+) tumors (do not derive benefit from TMZ treatment) are more likely to respond to sunitinib-based therapy. MGMT promoter methylation will be therefore used as a biomarker for selection of newly diagnosed GBM patients enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented newly diagnosed GBM patients
* Unmethylated MGMT promoter as determined by Methylation specific-polymerase chain reaction (MGMT(+) tumor)
* Age between 18 to 70
* Karnofsky performance status ≥70
* History and physical examination including neurologic examination within 4 weeks prior to registration
* Systolic blood pressure ≤ 160 mmHg or diastolic pressure ≤ 100mm Hg
* Required blood work within 14 days prior to registration
* Eligible for standard concurrent chemoradiation with TMZ
* Patients must have normal organ and marrow functions as defined below:

  * Absolute neutrophil count ≥ 1.5x 109/L
  * Platelets ≥100x 109/L
  * Hemoglobin ≥80g/L
  * International Normalized Ratio ≤1.3
  * Creatinine ≤1.5x [upper limit of normal] Or creatinine clearance ≥60 mL/min/1.73m2
* Normal baseline thyroid function as measured by a thyrotropic-stimulating hormone within institutional normal limits
* Adequate liver function: Alanine transaminase or Aspartate transaminase < 2 x upper limit of normal and bilirubin 1.6 mg/dL. No active bleeding or pathologic condition that carries high risk of bleeding (e.g. tumor involving major vessels or known varices)
* Patients who have undergone resection must meet the following conditions:

  * Patients must have recovered from the effects of surgery and a minimum of 14 to 28 days must have elapsed from the day of surgery to day of registration. Day of registration is considered the first day of Sunitinib.
  * For stereotactic biopsy, a minimum of 14 days must have elapsed prior to registration
* No prior RT to the brain, chemotherapy, or anti-angiogenic therapy
* Estimated life expectancy of at least 6 months
* Premenopausal women must have a negative human chorionic gonadotropin within 14 days prior to registration
* The effects of Sunitinib on the developing human fetus is unknown. Women of childbearing potential and male participants must practice adequate contraception. Should a woman become pregnant or suspect she is pregnant during the study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Histologically documented newly diagnosed GBM patients with methylated MGMT promoter
* Serious medical conditions that might be aggravated by treatment, including but not limited to: myocardial infarction within 6 months, congestive heart failure, unstable angina, active cardiomyopathy, unstable ventricular arrhythmia, uncontrolled hypertension, uncontrolled psychotic disorders, serious infections, active peptic ulcer disease, active liver disease or cerebrovascular disease with previous stroke
* Patients with a history of coagulopathy
* Evidence of intratumoural or peritumoural hemorrhage deemed significant by the treating physician
* ≥ 1+ proteinuria on two successive urine dipstick assessments
* thrombolytic therapy within 4 weeks
* Patient with prolonged of corrected QT interval of more than 450 msec in screening EKG will be excluded
* Women who are pregnant or nursing
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Sunitinib
* Previous treatment with Sunitinib or other inhibitors of the vascular endothelial growth factor signalling axis
* Bleeding disorders
* Concurrent use of anticoagulant or antiplatelet drugs
* Patients with any condition that impairs their ability to swallow Sunitinib (e.g. gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease).
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Sunitinib. In addition, these patients are at increased risk of lethal infections when treated with bone marrow-suppressive therapy
* Individuals with MRI non-compatible metal in the body, or unable to undergo MRI procedures.
* Allergy to gadolinium
* Patients with severe liver impairment will not be enrolled in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2012-08; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Tumor Response Rate | 24 weeks
  The primary endpoint of this study is tumor response rate and will be assessed using the Response Assessment in Neuro-Oncology criteria (RANO). Tumor response rate will be compared to standard of care in newly diagnosed Glioblastoma Multiforme.

SECONDARY OUTCOMES:
Overall Survival | at 6 month post treatment
Progression free survival | 6 months post treatment
Biomarkers (Cytokines) response | at 6 months post treatment
  PDGF, VEGF, sVEGF-R1 / R-2, basic fibroblast growth factor (bFGF), EGF, placental growth factor (PIGF), stromal cell-derived factor-1α (SDF-1), interleukin (IL) -1β, IL-6, IL-8, transforming growth factor α (TGF- α), angiopoietin 1 (Ang1), angiopoietin 2 (Ang2), and soluble Tek/Tie2 receptor (sTie2)
Adverse Events | Assessment of toxicity will continue until week 13 post-sunitinib
  Investigator will assess long-term tolerance/toxicity of Sunitinib-based therapy. Toxicity will be scored using NCI Clinical Trials Criteria for Adverse Events (CTCAE) Version 3.0 (http://ctep.info.nih.gov/).
level of functioning | at 6 months post treatment
  Will be measured using Eastern Cooperative Oncology Group (ECOG performance status) 0-5
Increase use of corticosteroids | at 6 months post treatment
  Increase in corticosteroid dosage by 50%; in the absence of other clinical explanations (such as pseudoprogression) may indicate tumour progression. Calling this evolution clinical tumour progression is at the investigator's discretion.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Tom Baker Cancer Center and University of Calgary, Calgary, Alberta
  - McGill University Health Centre, Montreal, Quebec

REFERENCES:
- [Background] Motzer RJ, Michaelson MD, Rosenberg J, Bukowski RM, Curti BD, George DJ, Hudes GR, Redman BG, Margolin KA, Wilding G. Sunitinib efficacy against advanced renal cell carcinoma. J Urol. 2007 Nov;178(5):1883-7. doi: 10.1016/j.juro.2007.07.030. Epub 2007 Sep 17. PMID 17868732
- [Background] Motzer RJ, Hutson TE, Tomczak P, Michaelson MD, Bukowski RM, Rixe O, Oudard S, Negrier S, Szczylik C, Kim ST, Chen I, Bycott PW, Baum CM, Figlin RA. Sunitinib versus interferon alfa in metastatic renal-cell carcinoma. N Engl J Med. 2007 Jan 11;356(2):115-24. doi: 10.1056/NEJMoa065044. PMID 17215529
- [Background] Motzer RJ, Bukowski RM. Targeted therapy for metastatic renal cell carcinoma. J Clin Oncol. 2006 Dec 10;24(35):5601-8. doi: 10.1200/JCO.2006.08.5415. PMID 17158546
- [Background] Motzer RJ, Rini BI, Bukowski RM, Curti BD, George DJ, Hudes GR, Redman BG, Margolin KA, Merchan JR, Wilding G, Ginsberg MS, Bacik J, Kim ST, Baum CM, Michaelson MD. Sunitinib in patients with metastatic renal cell carcinoma. JAMA. 2006 Jun 7;295(21):2516-24. doi: 10.1001/jama.295.21.2516. PMID 16757724
- [Background] Demetri GD, van Oosterom AT, Garrett CR, Blackstein ME, Shah MH, Verweij J, McArthur G, Judson IR, Heinrich MC, Morgan JA, Desai J, Fletcher CD, George S, Bello CL, Huang X, Baum CM, Casali PG. Efficacy and safety of sunitinib in patients with advanced gastrointestinal stromal tumour after failure of imatinib: a randomised controlled trial. Lancet. 2006 Oct 14;368(9544):1329-38. doi: 10.1016/S0140-6736(06)69446-4. PMID 17046465
- [Background] Faivre S, Delbaldo C, Vera K, Robert C, Lozahic S, Lassau N, Bello C, Deprimo S, Brega N, Massimini G, Armand JP, Scigalla P, Raymond E. Safety, pharmacokinetic, and antitumor activity of SU11248, a novel oral multitarget tyrosine kinase inhibitor, in patients with cancer. J Clin Oncol. 2006 Jan 1;24(1):25-35. doi: 10.1200/JCO.2005.02.2194. Epub 2005 Nov 28. PMID 16314617
- [Background] de Bouard S, Herlin P, Christensen JG, Lemoisson E, Gauduchon P, Raymond E, Guillamo JS. Antiangiogenic and anti-invasive effects of sunitinib on experimental human glioblastoma. Neuro Oncol. 2007 Oct;9(4):412-23. doi: 10.1215/15228517-2007-024. Epub 2007 Jul 10. PMID 17622648
- [Background] Abdollahi A, Lipson KE, Sckell A, Zieher H, Klenke F, Poerschke D, Roth A, Han X, Krix M, Bischof M, Hahnfeldt P, Grone HJ, Debus J, Hlatky L, Huber PE. Combined therapy with direct and indirect angiogenesis inhibition results in enhanced antiangiogenic and antitumor effects. Cancer Res. 2003 Dec 15;63(24):8890-8. PMID 14695206
- [Background] Frederick B, Gustafson D, Bianco C, Ciardiello F, Dimery I, Raben D. ZD6474, an inhibitor of VEGFR and EGFR tyrosine kinase activity in combination with radiotherapy. Int J Radiat Oncol Biol Phys. 2006 Jan 1;64(1):33-7. doi: 10.1016/j.ijrobp.2005.05.050. PMID 16377413
- [Background] Huber PE, Bischof M, Jenne J, Heiland S, Peschke P, Saffrich R, Grone HJ, Debus J, Lipson KE, Abdollahi A. Trimodal cancer treatment: beneficial effects of combined antiangiogenesis, radiation, and chemotherapy. Cancer Res. 2005 May 1;65(9):3643-55. doi: 10.1158/0008-5472.CAN-04-1668. PMID 15867359
- [Background] Schueneman AJ, Himmelfarb E, Geng L, Tan J, Donnelly E, Mendel D, McMahon G, Hallahan DE. SU11248 maintenance therapy prevents tumor regrowth after fractionated irradiation of murine tumor models. Cancer Res. 2003 Jul 15;63(14):4009-16. PMID 12873999
- [Background] Siemann DW, Rojiani AM. The vascular disrupting agent ZD6126 shows increased antitumor efficacy and enhanced radiation response in large, advanced tumors. Int J Radiat Oncol Biol Phys. 2005 Jul 1;62(3):846-53. doi: 10.1016/j.ijrobp.2005.02.048. PMID 15936569
- [Background] Chahal M, Xu Y, Lesniak D, Graham K, Famulski K, Christensen JG, Aghi M, Jacques A, Murray D, Sabri S, Abdulkarim B. MGMT modulates glioblastoma angiogenesis and response to the tyrosine kinase inhibitor sunitinib. Neuro Oncol. 2010 Aug;12(8):822-33. doi: 10.1093/neuonc/noq017. Epub 2010 Feb 23. PMID 20179017
- [Background] Bischof M, Abdollahi A, Gong P, Stoffregen C, Lipson KE, Debus JU, Weber KJ, Huber PE. Triple combination of irradiation, chemotherapy (pemetrexed), and VEGFR inhibition (SU5416) in human endothelial and tumor cells. Int J Radiat Oncol Biol Phys. 2004 Nov 15;60(4):1220-32. doi: 10.1016/j.ijrobp.2004.07.689. PMID 15519795